CLINICAL TRIAL: NCT01069419
Title: A Multicenter, Observational, Non-interventional Study to Evaluate the Safety and Efficacy of Anti-TNF (Anti-Tumor Necrosis Factor) Alpha Therapy With Certolizumab Pegol Observed in Daily Practice in Adult Rheumatoid Arthritis (RA) Patients
Brief Title: Observation of Treatment With Certolizumab Pegol in Daily Practice
Acronym: FasT
Status: Completed | Type: Observational
Sponsor: UCB Pharma GmbH (Industry)
Responsible Party: Sponsor
Organization: UCB Pharma (Industry)
Other Study IDs: RA0027
Record Dates: First submitted 2010-02-15; First posted 2010-02-17 (Estimated); Results first posted 2015-09-29 (Estimated); Last update posted 2015-10-29 (Estimated); Status verified 2015-10

CONDITIONS: Rheumatoid Arthritis
Keywords: Certolizumab Pegol; Cimzia
MeSH Terms: conditions — Arthritis, Rheumatoid

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Cimzia: All patients will be treated with Cimzia according to normal clinical practice for the prescribing physician and as defined by the SmPC

SUMMARY:
This is an observational, non-interventional, non-comparative, post-authorization safety study to evaluate efficacy and long-term safety of Cimzia in adult patients with RA in need of treatment with a biological product.

DETAILED DESCRIPTION:
The purpose of this study is to assess the clinical efficacy of Cimzia in achieving clinical remission after two years of therapy. The observational nature of the study leaves the therapeutic decision exclusively within the discretion of the treating physician.

ELIGIBILITY:
Inclusion Criteria:

* Patients eligible for treatment with Cimzia as defined in EU approved SmPC

Exclusion Criteria:

* Patient previously treated with Cimzia. Patient with known hypersensitivity to any component of Cimzia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Male or female ≥ 18 years of age with RA and is eligible for treatment with Cimzia. Recruited in Germany.
Sampling Method: Non-Probability Sample
Enrollment: 1117 (Actual)
Dates: Start 2009-10; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: UCB Clinical Trial Call center, Study Director — +1 877 822 9493 (UCB)
Locations (163):
- Germany (163):
  - 174, Altenburg
  - 70, Amberg
  - 122, Attendorn
  - 153, Augsburg
  - 3, Bad Aibling
  - 133, Bad Bramstedt
  - 167, Bad Buchau
  - 20, Bad Doberan
  - 166, Bad Endbach
  - 8, Bad Iburg
  - 66, Bad Kissingen
  - 137, Bad Kreuznach
  - 119, Bad Liebenwerda
  - 4, Bad Nauheim
  - 13, Bad Neuenahr-Ahrweiler
  - 87, Bad Staffelstein
  - 173, Baden-Baden
  - 19, Bamberg
  - 115, Bautzen
  - 21, Bayreuth
  - 58, Bayreuth
  - 112, Berlin
  - 12, Berlin
  - 163, Berlin
  - 179, Berlin
  - 1, Berlin
  - 25, Berlin
  - 26, Berlin
  - 43, Berlin
  - 54, Berlin
  - 59, Berlin
  - 61, Berlin
  - 72, Berlin
  - 78, Berlin
  - 91, Berlin
  - 95, Berlin
  - 28, Chemnitz
  - 75, Chemnitz
  - 16, Cologne
  - 73, Cologne
  - 97, Cologne
  - 134, Darmstadt
  - 71, Darmstadt
  - 125, Deggendorf
  - 131, Dresden
  - 36, Dresden
  - 88, Dresden
  - 98, Dresden
  - 49, Duisburg
  - 46, Düsseldorf
  - 102, Elmshorn
  - 83, Erfurt
  - 2, Erlangen
  - 37, Essen
  - 84, Essen
  - 136, Frankenberg-Sachsen
  - 103, Frankfurt
  - 53, Frankfurt
  - 29, Freiberg
  - 86, Freiburg im Breisgau
  - 77, Fulda
  - 15, Goslar
  - 100, Göttingen
  - 89, Gräfelfing
  - 135, Greifswald
  - 107, Güstrow
  - 157, Hagen
  - 150, Haldensleben I
  - 11, Halle
  - 116, Hamburg
  - 128, Hamburg
  - 139, Hamburg
  - 175, Hamburg
  - 50, Hamburg
  - 55, Hamburg
  - 67, Hamburg
  - 6, Hamburg
  - 129, Hanau
  - 159, Hanover
  - 171, Hanover
  - 17, Hanover
  - 138, Heidelberg
  - 146, Heidelberg
  - 47, Heidelberg
  - 92, Heilbad Heiligenstadt
  - 64, Herrsching am Ammersee
  - 5, Hildesheim
  - 30, Hofheim
  - 48, Hoyerswerda
  - 130, Karlsruhe
  - 56, Karlsruhe
  - 96, Karlsruhe
  - 101, Karlstadt am Main
  - 121, Kassel
  - 161, Katzhütte
  - 158, Kiel
  - 127, Leipzig
  - 51, Ludwigsfelde
  - 140, Ludwigslust
  - 93, Lübeck
  - 68, Magdeburg
  - 145, Mainz
  - 31, Marktredwitz
  - 94, Mittelherwigsdorf
  - 18, Mönchengladbach
  - 104, Mühlheim An Der Ruhr
  - 10, München
  - 164, München
  - 178, München
  - 9, München
  - 113, Münster
  - 123, Münster
  - 57, Naunhof
  - 32, Neubrandenburg
  - 108, Neuburg am Inn
  - 149, Neuruppin
  - 44, Neuss
  - 7, Nienburg
  - 141, Norderstedt
  - 172, Nuremberg
  - 22, Nuremberg
  - 99, Oberammergau
  - 23, Oberhausen
  - 33, Offenburg
  - 38, Osnabrück
  - 154, Paderborn
  - 34, Pirna
  - 81, Planegg
  - 85, Plauen
  - 27, Potsdam
  - 35, Potsdam
  - 24, Ratingen
  - 82, Rendsburg
  - 124, Rheine
  - 109, Rostock
  - 76, Rostock
  - 90, Rüdersdorf
  - 39, Saarbrücken
  - 69, Salzwedel
  - 117, Schramberg-Sulgen
  - 143, Schwerin
  - 142, Schwerte
  - 120, Seesen
  - 105, Stadtbergen
  - 14, Stuttgart
  - 40, Stuttgart
  - 160, Traunstein
  - 170, Treuenbrietzen
  - 41, Tübingen
  - 168, Uffenheim
  - 111, Ulm
  - 65, Ulm
  - 52, Villingen-Schwenningen
  - 106, Weener
  - 162, Weiden
  - 177, Weißenfels
  - 118, Wiesbaden
  - 74, Wiesbaden
  - 60, Winsen
  - 165, Würselen
  - 152, Würzburg
  - 110, Zeven
  - 45, Zwiesel

REFERENCES:
- See also: FDA Safety Alerts and Recalls — http://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This non-interventional study started to enroll participants in Germany in October 2009 and concluded in December 2014.
  Participant Flow refers to the Enrolled Set.
Pre-assignment Details: There were 13 patients with missing termination information. Therefore only safety data were analyzed for these 13 patients. Patients with missing termination information were neither considered as completer nor as non-completer in the Clinical Study Report. These patients are considered as non-completers in the summary below.
Period: Overall Study
Arm/Group | Cimzia
Started | 1117
Safety Set | 1111
Full Analysis Set | 851
Completed | 402
Not Completed | 715
Not completed — Adverse Event | 233
Not completed — Lack of Efficacy | 332
Not completed — Lost to Follow-up | 49
Not completed — Remission of disease | 11
Not completed — Withdrawal by Subject | 34
Not completed — Other Reason | 43
Not completed — Missing termination information | 13

BASELINE CHARACTERISTICS:
Population: Baseline Characteristics refer to the Enrolled Set.
Arm/Group | Cimzia
Number analyzed (Participants) | 1117
Age, Customized [Number; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 848
  >=65 years | 268
  Missing | 1
Age, Continuous [Mean (Standard Deviation); unit: years] — One subject's age data was missing. Age continuous calculation is based on n=1116.
  years | 55.1 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 870
  Male | 247

OUTCOME MEASURES:

1. Primary Outcome: Clinical Remission at Visit 9 (Around Week 104) Measured by Achieving a Disease Activity Score 28 (DAS28) of < 2.6
Description: The DAS28 was calculated using the tender and swollen joint counts, c-reactive Protein (CRP), or erythrocyte sedimentation rate (ESR), and the Patient's Global Assessment of Disease Activity (PtGADA). The joint assessment was carried out on 28 joints.
  For the analysis, DAS28 values were categorized into the following groups:
  * DAS28 < 2.6: clinical remission
  * DAS28 from 2.6 to ≤ 3.2: low disease activity
  * DAS28 from > 3.2 to 5.1: moderate disease activity
  * DAS28 > 5.1: high disease activity
Time Frame: From Baseline to Visit 9 (around Week 104)
Population: Full Analysis Set (FAS) using Non-Responder Imputation (NRI). FAS is defined as all patients with a DAS28 ≥ 2.6 at baseline who took at least 1 dose of Certolizumab Pegol and had at least 1 valid post-Baseline DAS28 value.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Cimzia
Number analyzed (Participants) | 851
percentage of participants | 14.1 [11.8 to 16.4]

2. Secondary Outcome: Change From Baseline to Visit 9 (Around Week 104) in Patients's Arthritis Pain as Measured by Patient's Assessment of Arthritis Pain (PAAP) Visual Analog Scale (VAS)
Description: Patients rated how much pain they were experiencing at the time of the visit caused by their Arthritis using a Visual Analog Scale (VAS) ranging from 0 (no pain) to 100 (most severe pain). A negative value in Change from Baseline indicates an improvement from Baseline to Visit 9 (around Week 104).
Time Frame: From Baseline to Visit 9 (around Week 104)
Population: Full Analysis Set (FAS) using Mixed Model with Repeated Measures imputation (MMRM). FAS is defined as all patients with a DAS28 ≥ 2.6 at baseline who took at least 1 dose of Certolizumab Pegol and had at least 1 valid post-Baseline DAS28 value.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cimzia
Number analyzed (Participants) | 845
units on a scale | -16.43 (20.34)

3. Secondary Outcome: Change From Baseline to Visit 9 (Around Week 104) in Patient's Physical Function as Measured by the Health Assessment Questionnaire-Disability Index (HAQ-DI)
Description: The HAQ-DI contains 20 items on a 4-point scale ranging from 0 (without any difficulty) to 3 (unable to do). The 20 items are grouped in 8 categories with 2 to 3 items each. The category scores are averaged into an overall HAQ-DI from 0 to 3. Scores of 0 to 1 generally represent mild to moderate difficulty, 1 to 2 represent moderate to severe disability, and 2 to 3 indicate severe to very severe disability. A negative value in Change from Baseline indicates an improvement from Baseline to Visit 9 (around Week 104).
Time Frame: From Baseline to Visit 9 (around Week 104)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cimzia
Number analyzed (Participants) | 845
units on a scale | -0.26 (0.39)

4. Secondary Outcome: Change From Baseline to Visit 9 (Around Week 104) in Disease Activity Measured by Clinical Disease Activity Index (CDAI)
Description: The CDAI was calculated with the equation:
  CDAI= Tender Joint Count + Swollen Joint Count + PtGADA/10 + PhGADA/10 where PtGADA (mm) is the Patient's Global Assessment of Disease Activity using a Visual Analog Scale (VAS) ranging from 0 to 100, and PhGADA (mm) is the Physician's Global Assessment of Disease Activity using a VAS ranging from 0 to 100. Thus, the CDAI ranges from 0 to 76, with higher values indicating higher disease activity. If any individual term was missing, then the CDAI was set to missing. A negative value in Change from Baseline indicates an improvement from Baseline to Visit 9 (around Week 104).
Time Frame: From Baseline to Visit 9 (around Week 104)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Cimzia
Number analyzed (Participants) | 846
units on a scale | -14.57 (10.24)

ADVERSE EVENTS:
Time Frame: Adverse Events were collected from Visit 2 (Week 6) up to Visit 10 (Week 116).
Description: Adverse Events refer to the Safety Set consisting of all enrolled subjects who took at least one dose of Certolizumab Pegol.
Arm/Group | Cimzia
Serious Adverse Events (participants affected / at risk) | 212/1111
Other Adverse Events (participants affected / at risk) | 111/1111
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cimzia (N=1111)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (1)
Anaemia (Blood and lymphatic system disorders) | 2 (2)
Leukocytosis (Blood and lymphatic system disorders) | 1 (1)
Lymphadenitis (Blood and lymphatic system disorders) | 1 (1)
Thrombocytopenia (Blood and lymphatic system disorders) | 1 (1)
Cardiovascular insufficiency (Cardiac disorders) | 1 (1)
Coronary artery disease (Cardiac disorders) | 4 (4)
Cardiac failure chronic (Cardiac disorders) | 3 (3)
Cardiac failure (Cardiac disorders) | 2 (3)
Myocardial infarction (Cardiac disorders) | 2 (2)
Acute myocardial infarction (Cardiac disorders) | 1 (1)
Dilatation ventricular (Cardiac disorders) | 1 (1)
Arrhythmia (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Tachycardia (Cardiac disorders) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 2 (2)
Sinus tachycardia (Cardiac disorders) | 1 (1)
Supraventricular tachycardia (Cardiac disorders) | 1 (1)
Ventricular fibrillation (Cardiac disorders) | 1 (1)
Hyperthyroidism (Endocrine disorders) | 1 (2)
Cataract (Eye disorders) | 1 (1)
Iridocyclitis (Eye disorders) | 1 (2)
Retinal artery occlusion (Eye disorders) | 1 (1)
Retinal detachment (Eye disorders) | 1 (1)
Colitis ischaemic (Gastrointestinal disorders) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 2 (2)
Diarrhoea haemorrhagic (Gastrointestinal disorders) | 1 (1)
Diverticulum intestinal (Gastrointestinal disorders) | 1 (1)
Duodenal ulcer (Gastrointestinal disorders) | 1 (1)
Gastric ulcer perforation (Gastrointestinal disorders) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 1 (1)
Mechanical ileus (Gastrointestinal disorders) | 1 (1)
Large intestine perforation (Gastrointestinal disorders) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (2)
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Melaena (Gastrointestinal disorders) | 1 (1)
Ascites (Gastrointestinal disorders) | 1 (1)
Parotid gland enlargement (Gastrointestinal disorders) | 1 (1)
Umbilical hernia (Gastrointestinal disorders) | 1 (1)
Death (General disorders) | 1 (1)
Unevaluable event (General disorders) | 2 (2)
Local swelling (General disorders) | 1 (1)
Chest pain (General disorders) | 1 (1)
Drug intolerance (General disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Cholelithiasis (Hepatobiliary disorders) | 1 (1)
Autoimmune hepatitis (Hepatobiliary disorders) | 1 (1)
Hypersensitivity (Immune system disorders) | 1 (1)
Anaphylactic reaction (Immune system disorders) | 1 (1)
Diverticulitis (Infections and infestations) | 2 (2)
Gastroenteritis (Infections and infestations) | 1 (1)
Gastrointestinal infection (Infections and infestations) | 1 (1)
Peritonitis (Infections and infestations) | 1 (1)
Arthritis bacterial (Infections and infestations) | 1 (1)
Cellulitis (Infections and infestations) | 1 (1)
Cellulitis gangrenous (Infections and infestations) | 1 (1)
Mastitis (Infections and infestations) | 1 (1)
Cystitis escherichia (Infections and infestations) | 1 (1)
Escherichia sepsis (Infections and infestations) | 1 (1)
Gallbladder empyema (Infections and infestations) | 1 (1)
Liver abscess (Infections and infestations) | 1 (1)
Herpes zoster (Infections and infestations) | 1 (1)
Ophthalmic herpes zoster (Infections and infestations) | 1 (1)
Abscess (Infections and infestations) | 1 (1)
Abscess limb (Infections and infestations) | 1 (1)
Localised infection (Infections and infestations) | 1 (1)
Postoperative wound infection (Infections and infestations) | 1 (1)
Influenza (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 10 (10)
Bronchopneumonia (Infections and infestations) | 2 (2)
Bronchitis (Infections and infestations) | 1 (1)
Epididymitis (Infections and infestations) | 1 (1)
Muscle abscess (Infections and infestations) | 1 (1)
Sepsis (Infections and infestations) | 4 (4)
Erysipelas (Infections and infestations) | 2 (2)
Pneumonia pneumococcal (Infections and infestations) | 1 (1)
Pulmonary tuberculosis (Infections and infestations) | 2 (2)
Tuberculosis (Infections and infestations) | 2 (2)
Urinary tract infection (Infections and infestations) | 3 (4)
Cystitis (Infections and infestations) | 1 (1)
Gastrointestinal viral infection (Infections and infestations) | 1 (1)
Viral infection (Infections and infestations) | 1 (1)
Post procedural myocardial infarction (Injury, poisoning and procedural complications) | 1 (1)
Craniocerebral injury (Injury, poisoning and procedural complications) | 1 (1)
Joint dislocation (Injury, poisoning and procedural complications) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 2 (2)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2)
Femur fracture (Injury, poisoning and procedural complications) | 1 (1)
Tibia fracture (Injury, poisoning and procedural complications) | 1 (1)
Tendon rupture (Injury, poisoning and procedural complications) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 1 (1)
Multiple injuries (Injury, poisoning and procedural complications) | 1 (1)
Injection related reaction (Injury, poisoning and procedural complications) | 1 (1)
Pelvic fracture (Injury, poisoning and procedural complications) | 1 (1)
Contusion (Injury, poisoning and procedural complications) | 1 (1)
Skull fracture (Injury, poisoning and procedural complications) | 1 (1)
Dislocation of vertebra (Injury, poisoning and procedural complications) | 1 (1)
Forearm fracture (Injury, poisoning and procedural complications) | 2 (2)
Humerus fracture (Injury, poisoning and procedural complications) | 1 (2)
Anti-cyclic citrullinated peptide antibody positive (Investigations) | 1 (1)
Liver function test abnormal (Investigations) | 1 (1)
Blood pressure increased (Investigations) | 1 (1)
Type 2 diabetes mellitus (Metabolism and nutrition disorders) | 2 (2)
Diabetes mellitus (Metabolism and nutrition disorders) | 1 (1)
Gout (Metabolism and nutrition disorders) | 1 (1)
Arthritis (Musculoskeletal and connective tissue disorders) | 3 (3)
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Bone infarction (Musculoskeletal and connective tissue disorders) | 1 (3)
Osteonecrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal disorder (Musculoskeletal and connective tissue disorders) | 1 (1)
Bursitis (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteochondrosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Foot deformity (Musculoskeletal and connective tissue disorders) | 3 (3)
Wrist deformity (Musculoskeletal and connective tissue disorders) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 3 (3)
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 2 (2)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoporosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 (1)
Spinal pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 (7)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 22 (23)
Felty's syndrome (Musculoskeletal and connective tissue disorders) | 1 (1)
Rheumatoid nodule (Musculoskeletal and connective tissue disorders) | 1 (1)
Neck mass (Musculoskeletal and connective tissue disorders) | 1 (1)
Lumbar spinal stenosis (Musculoskeletal and connective tissue disorders) | 2 (2)
Spinal column stenosis (Musculoskeletal and connective tissue disorders) | 1 (1)
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1 (1)
Synovitis (Musculoskeletal and connective tissue disorders) | 5 (8)
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cervix carcinoma stage 0 (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Benign salivary gland neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Metastases to central nervous system (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Ovarian germ cell teratoma benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Bronchial carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Small cell lung cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Thyroid cancer recurrent (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 2 (2)
Cerebral infarction (Nervous system disorders) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Ischaemic cerebral infarction (Nervous system disorders) | 1 (1)
Syncope (Nervous system disorders) | 1 (1)
Facial paresis (Nervous system disorders) | 1 (1)
Generalised tonic-clonic seizure (Nervous system disorders) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 2 (2)
Paraesthesia (Nervous system disorders) | 1 (1)
Hemiparesis (Nervous system disorders) | 1 (1)
Paralysis flaccid (Nervous system disorders) | 1 (1)
Transient ischaemic attack (Nervous system disorders) | 4 (4)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1)
Depression (Psychiatric disorders) | 2 (2)
Schizoaffective disorder depressive type (Psychiatric disorders) | 1 (1)
Acute prerenal failure (Renal and urinary disorders) | 1 (1)
Renal failure (Renal and urinary disorders) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1)
Nephrolithiasis (Renal and urinary disorders) | 2 (2)
Urethral polyp (Renal and urinary disorders) | 1 (1)
Ovarian mass (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Vocal cord cyst (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleurisy (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Dermatitis allergic (Skin and subcutaneous tissue disorders) | 3 (3)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema (Skin and subcutaneous tissue disorders) | 1 (1)
Erythema nodosum (Skin and subcutaneous tissue disorders) | 1 (1)
Psoriasis (Skin and subcutaneous tissue disorders) | 4 (4)
Pustular psoriasis (Skin and subcutaneous tissue disorders) | 2 (2)
Dermatitis psoriasiform (Skin and subcutaneous tissue disorders) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 1 (1)
Rash vesicular (Skin and subcutaneous tissue disorders) | 1 (1)
Analgesic therapy (Surgical and medical procedures) | 1 (1)
Synovectomy (Surgical and medical procedures) | 3 (3)
Knee arthroplasty (Surgical and medical procedures) | 2 (2)
Polypectomy (Surgical and medical procedures) | 1 (2)
Hypertensive crisis (Vascular disorders) | 2 (2)
Haematoma (Vascular disorders) | 1 (1)
Deep vein thrombosis (Vascular disorders) | 4 (4)
Varicophlebitis (Vascular disorders) | 1 (1)
Hypertension (Vascular disorders) | 3 (3)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cimzia (N=1111)
Nasopharyngitis (Infections and infestations) | 111 (143)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days